CLINICAL TRIAL: NCT07346781
Title: Effects of Social Cognitive Theory-Based Eco-Friendly Nutrition Education on Sustainable Food Literacy and Nutritional Behaviors in Women: A Randomized Controlled Trial
Brief Title: Effects of Eco-Friendly Nutrition Education on Sustainable Food Literacy and Nutritional Behaviors in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sumeyra YILMAZ, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: E-77082166-604.01-1217558
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-05

CONDITIONS: Sustainable Healthy Diet; Food Literacy
Keywords: sustainable health nutrition; women; food literacy; public health

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: To prevent selection bias in the study, adolescents were randomly assigned to the intervention and control groups by an independent biostatistician using a simple randomization method. Participant numbers were assigned when the preliminary assessment data were transferred to the computer. The researcher was unaware of the participants' group status until the study began. The data were coded and transferred to the computer without specifying the intervention and control groups. To prevent reporting bias, the study data were evaluated by an independent biostatistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eco-Friendly Nutrition Educational Intervention Group (Experimental): The intervention program was created in five sessions based on a comprehensive literature review and Social Cognitive Theory to improve women's sustainable food literacy and sustainable nutritional behaviors. After each topic is presented by the researcher, various interactive practices such as reviewing reliable websites on the topic, reviewing food packages, reviewing brochures prepared by the researcher will be included to improve food literacy and sustainable nutritional behaviors and gain critical evaluation skills. The intervention sessions will be held in a room approved by the institution administration in the Women's Club. The intervention sessions will be held in five sessions, each approximately 45 minutes long, at one-week intervals. In order to organize the intervention sessions, the participating women will be contacted by phone and a suitable date and time will be determined. The planned time will be reminded by text message on the day of the intervention session. In or
  Interventions: Behavioral: Eco-Friendly Nutrition Educational Intervention Program
- Waiting List Control Group (Other): No intervention will be made to the women in the waiting list group during the intervention group training process and the research process. After the completion of the training process of the women in the intervention group and the post-test data and the follow-up test one month later, the interventions will be applied to
  Interventions: Behavioral: Eco-Friendly Nutrition Educational Intervention Program

INTERVENTIONS:
Behavioral: Eco-Friendly Nutrition Educational Intervention Program — The intervention sessions will be held in a room approved by the institution administration in the Women's Club. The intervention sessions will be held in five sessions, each approximately 45 minutes long, at one-week intervals. In order to organize the intervention sessions, the participating women will be contacted by phone and a suitable date and time will be determined. The planned time will be reminded by text message on the day of the intervention session. In order to prevent loss and ensure that the intervention sessions continue as group training, participants who cannot attend the planned session will be included in another group addressing the same topic.

SUMMARY:
This research will be conducted face-to-face with women registered at the Women's Club. Participants included in the study are expected to fill out three survey forms first. The first form includes the Descriptive Information Form, which includes questions such as age, height, weight, marital status, education, employment status, and income status; the second form includes the Food Literacy Tool; and the third form includes the Behavior Scale for Sustainable Nutrition. It takes approximately 20 minutes to fill out the forms. After the survey forms are filled out, participants will be randomly divided into two groups and the order of the groups will be determined by drawing lots. Participants in the first group will attend the Environmentally Friendly Nutrition Training once a week for five weeks immediately after the survey forms are filled out. Participants in the second group will be included in the training after the first group's training is completed. The survey form will be filled out again immediately after the training and one month later. The study will be completed with the completion of the last surveys.

DETAILED DESCRIPTION:
This research will be conducted face-to-face with women registered at the Women's Club. Participants included in the study are expected to fill out three survey forms first. The first form includes the Descriptive Information Form, which includes questions such as age, height, weight, marital status, education, employment status, and income status; the second form includes the Food Literacy Tool; and the third form includes the Behavior Scale for Sustainable Nutrition. It takes approximately 20 minutes to fill out the forms. After the survey forms are filled out, participants will be randomly divided into two groups and the order of the groups will be determined by drawing lots. Participants in the first group will attend the Environmentally Friendly Nutrition Training once a week for five weeks immediately after the survey forms are filled out. The training is based on Social Cognitive Theory. Each week is designed with various practices and activities in addition to theoretical training. Participants assigned to the second group will be included in the training after the first group's training is completed. The survey form will be filled out again immediately after the training and one month later. The study will be completed with the completion of the last surveys.

ELIGIBILITY:
Inclusion Criteria:

* Being registered with the municipality's Women's Club, Participating in the study voluntarily, not having a language barrier in communication and not having received training on environmentally friendly nutrition before.

Exclusion Criteria:

* not meeting inclusion criteria

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Responsibilities such as shopping for the necessary ingredients for meals, preparation, cooking, gardening, and removing food waste from the home are generally undertaken by women. Therefore, it is important to determine women's food literacy and sustainable environmentally friendly nutritional behaviors. Therefore, this research includes women in the sample.
Enrollment: 122 (Actual)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-06-04 (Actual); Study Completion 2025-09-04 (Actual)

PRIMARY OUTCOMES:
Sustainable Food Literacy Tool Score | before intervention (week 1)after intervention (week 5)follow-up time (at the end of the 3rd month)
  The Turkish validity and reliability of the scale developed by Rosas et al. (2022) was made by Ertaş Öztürk et al. (2024). The scale contains 24 items, five factors (F1: Culinary competencies, F2: Production and quality, F3: Selection and planning, F4: Environmentally safe, F5: Origin) and a Likert-type scoring system (0-never/completely disagree, 1-sometimes/disagree, 2-often/agree, 3-always/completely agree). Each item is scored between 0 and 3 points. The total score and the scores of the sub-factors are obtained by summing up the relevant items. The score obtained shows the level of sustainable food literacy. The Cronbach alpha internal consistency coefficient of the entire scale is 0.831.
General Self-Efficacy Scale Score | before intervention (week 1)after intervention (week 5)follow-up time (at the end of the 3rd month)
  General Self-Efficacy Scale The Turkish validity and reliability of the scale developed by Sherer et al. (1982) was carried out by Yıldırım and İlhan (2010). The scale consists of 17 items and three sub-dimensions (Initiation, Not Giving Up, Sustainment Effort-Persistence). It has a Likert-type five-point rating from not at all to very good, and items 2, 4, 5, 6, 7, 10, 11, 12, 14, 16 and 17 are reverse scored. The total score of the scale can vary between 17-85. An increase in the total score indicates an increase in self-efficacy belief. The Cronbach alpha internal consistency coefficient of the entire scale was found to be 0.80.
Sustainable Nutrition Behavior Scale Score | before intervention (week 1)after intervention (week 5)follow-up time (at the end of the 3rd month)
  Sustainable Nutrition Behavior Scale Developed by Garipoglu et al. (2023). It consists of 29 items and 4 sub-dimensions (food preference, reduction of food waste, seasonal and local nutrition, purchasing food) with a five-point Likert-type scale. The scale is rated as "never", "rarely", "sometimes", "often" and "always". All items are scored from 1 to 5, starting from the "never" option. The lowest score that can be obtained from the scale is 29 and the highest score is 145. Sub-dimension scores are obtained by dividing the sum of the scores given by individuals to the questions in the sub-dimension by the number of questions in the sub-dimension. Higher total scores and sub-dimension scores indicate that the individual has more sustainable nutrition behaviors. The Cronbach alpha internal consistency coefficient of the entire scale was found to be 0.92.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Metropolitan Municipality, Ladies' Club, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
In order to protect the personal information of the participants, their data is not shared. However, the authors can be contacted for explainable reasons.